CLINICAL TRIAL: NCT07070661
Title: Effects of Radial Pressure Wave Therapy Modulation in Patients With Carpal Tunnel Syndrome: A Double-Blind Randomized Clinical Trial.
Brief Title: Radial Pressure Wave Therapy With or Without Parameter Modulation for Carpal Tunnel Syndrome.
Acronym: RPWT in CTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armando Tonatiuh Avila Garcia (Other)
Collaborators: University of Guadalajara (Other)
Responsible Party: Sponsor-Investigator, Armando Tonatiuh Avila Garcia, Chief Department of Physical Medicine and Rehabilitation, Hospital Civil de Guadalajara
Organization: Hospital Civil de Guadalajara (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI 144/25
Record Dates: First submitted 2025-06-27; First posted 2025-07-17 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome; Radial Pressure Wave Therapy; Extracorporeal Shock Wave Therapy; Median Nerve; Neuropathic Pain; Hand Function; Non-invasive Treatment; Physical Medicine and Rehabilitation; Electrophysiology; Grip Strength
MeSH Terms: conditions — Carpal Tunnel Syndrome; Neuralgia

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial with two parallel groups comparing constant-dose versus modulated-dose radial pressure wave therapy in patients with carpal tunnel syndrome.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors (including the specialists in rehabilitation and neurophysiology) are blinded to group allocation. The intervention is applied by a therapist aware of the group assignment, but not involved in the evaluation or data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed-Dose Radial Pressure Wave Therapy. (Experimental): Participants assigned to this group will receive radial pressure wave therapy using a standardized protocol with fixed parameters of frequency and pressure throughout each session. The treatment will be administered once a week for three consecutive weeks. This group serves as the reference condition for comparative purposes.
  Interventions: Device: Fixed-Dose Radial Pressure Wave Therapy.
- Modulated-Dose Radial Pressure Wave Therapy. (Experimental): Participants in this group will receive radial pressure wave therapy with dynamic modulation of frequency and pressure during each session. The modulation will follow a predefined progressive scheme aimed at optimizing tissue response. Treatment will be delivered once a week for three consecutive weeks.
  Interventions: Device: Modulated-Dose Radial Pressure Wave Therapy.

INTERVENTIONS:
Device: Fixed-Dose Radial Pressure Wave Therapy. — Radial pressure wave therapy will be delivered using the BTL-6000 device. Parameters such as frequency and pressure will remain constant throughout each session. Each participant will receive one session per week for three weeks. The treatment will follow a standardized protocol previously established in the literature and based on patient tolerance.
  Arms: Fixed-Dose Radial Pressure Wave Therapy.
Device: Modulated-Dose Radial Pressure Wave Therapy. — The BTL-6000 device will be used to deliver therapy with dynamic modulation of frequency and/or pressure within each session, following a structured protocol aiming to optimize clinical response.
  Arms: Modulated-Dose Radial Pressure Wave Therapy.

SUMMARY:
This study aims to evaluate the clinical effects of radial pressure wave therapy in patients with a confirmed diagnosis of mild to moderate carpal tunnel syndrome. Participants will be randomly assigned to receive radial pressure wave therapy using either a modulated or a constant parameter dosing protocol. The intervention consists of three weekly sessions, and outcomes will be assessed at baseline, 2 months, and 4 months after the first session. The primary outcome is pain intensity measured by the Visual Analog Scale, while secondary outcomes include functional status evaluated with the Boston Carpal Tunnel Questionnaire, grip strength, and electrodiagnostic parameters of the median nerve. The study is conducted in the Physical Medicine and Rehabilitation Service of the Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde," and has been approved by the hospital's Ethics Committee.

DETAILED DESCRIPTION:
This is a double-blind randomized controlled trial designed to explore the effects of different dosing strategies of radial pressure wave therapy in patients with mild to moderate carpal tunnel syndrome. Sixty patients aged 18 to 75 years, with clinical and electrodiagnostic confirmation of CTS, will be recruited and randomly assigned (1:1) to one of two intervention groups: (1) RPWT with constant parameters; or (2) RPWT with modulated parameters (progressive variation of frequency and pressure during each session). All participants will receive three weekly sessions of RPWT and follow a standardized home-based exercise protocol for wrist and hand mobility.

The primary outcome will be the change in pain intensity, measured with the Visual Analog Scale VAS. Secondary outcomes include functional status assessed with the Boston Carpal Tunnel Questionnaire, grip strength using a calibrated hydraulic hand dynamometer, and neurophysiological parameters such as sensory conduction velocity, distal motor latency, and CMAP amplitude of the median nerve. Neurophysiological evaluations will be performed using the Nicolet Viking Quest system following standardized protocols.

Assessments will take place at baseline, 2 months, and 4 months after treatment initiation, except for electrodiagnostic studies which will be performed only at baseline and at 4 months. Statistical analysis will include mixed-design repeated measures ANOVA to assess intra- and inter-group effects and time-by-group interactions. The study complies with ethical standards and good clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* Clinical diagnosis of carpal tunnel syndrome based on symptoms such as nocturnal paresthesia, numbness in the median nerve distribution, and/or thenar weakness.
* At least one positive provocative test (e.g., Tinel's, Phalen's, or Durkan's test).
* Symptoms present for at least 1 month.
* NPRS (Numeric Pain Rating Scale) score ≥ 4 at baseline.
* Able and willing to attend all intervention sessions and follow-up assessments.
* Able to provide informed consent.

Exclusion Criteria:

* Prior wrist surgery on the affected side.
* Prior treatment with radial pressure wave therapy for CTS.
* Diagnosis of polyneuropathy, cervical radiculopathy, or systemic conditions affecting nerve function (e.g., uncontrolled diabetes, hypothyroidism, rheumatoid arthritis).
* Severe thenar atrophy or muscle wasting.
* Pacemaker or other implanted electronic devices.
* Pregnancy.
* Currently participating in another clinical trial or intervention study.
* Inability to understand or complete the study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured with the Numeric Pain Rating Scale. | Baseline, 2 months, and 4 months after treatment initiation.
  Pain intensity will be assessed using the 11-point Numeric Pain Rating Scale (0 = no pain, 10 = worst imaginable pain). The primary endpoint is the change in Numeric Pain Rating Scale score from baseline to the follow-up visits.

SECONDARY OUTCOMES:
Change in Self-Reported Function Using the Boston Carpal Tunnel Questionnaire. | Baseline, 2 months, and 4 months after treatment initiation.
  Function will be evaluated with the Functional Status Scale of the Boston Carpal Tunnel Questionnaire, which includes 8 items rated from 1 (no difficulty) to 5 (cannot perform activity). The mean score will be analyzed.
Grip strength measured with hydraulic hand dynamometer. | Baseline, 2 months, and 4 months after the first treatment session.
  Grip strength will be assessed using a calibrated Baseline® hydraulic hand dynamometer (range: 0-100 kg), following the standardized protocol recommended by the American Society of Hand Therapists. Patients will be seated with the shoulder adducted and neutrally rotated, elbow flexed at 90°, forearm in neutral position, and wrist in slight extension. Each participant will perform three maximal grip attempts, with brief rest periods in between, and the highest value will be recorded for analysis.
Change in Distal Motor Latency of the Median Nerve. | Baseline and 4 months after the first treatment session.
  Distal motor latency of the median nerve will be assessed using standard nerve conduction study protocols with surface electrodes and supramaximal stimulation. Values will be recorded in milliseconds, and the change from baseline to follow-up will be analyzed.
Change in Compound Muscle Action Potential (CMAP) Amplitude of the Median Nerve. | Baseline and 4 months after the first treatment session.
  CMAP amplitude will be measured from the median nerve using a standard supramaximal stimulation protocol and recorded in millivolts. The change in peak amplitude between baseline and follow-up will be used for analysis.
Change in Motor Nerve Conduction Velocity of the Median Nerve. | Baseline and 4 months after the first treatment session.
  Median motor nerve conduction velocity will be assessed using standard nerve conduction studies and calculated in meters per second. The highest conduction velocity from each assessment will be considered for analysis.
Change in Sensory Nerve Latency of the Median Nerve. | Baseline and 4 months after the first treatment session.
  Latency of the sensory action potential in the median nerve will be measured using standard antidromic stimulation techniques and recorded in milliseconds. The change from baseline to follow-up will be analyzed.
Change in Sensory Nerve Action Potential (SNAP) Amplitude of the Median Nerve. | Baseline and 4 months after the first treatment session.
  SNAP amplitude of the median nerve will be recorded using standard protocols and expressed in microvolts. The highest amplitude obtained will be compared between baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Tonatiuh Avila, MD, Principal Investigator — Hospital Civil de Guadalajara
Locations (1):
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the findings of this study are available from the lead author upon reasonable request by email.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From February 2026 to February 2027.
Access Criteria: 1. Qualified researchers who have received IRB approval.
  2. Prior reasonable request by email.
  3. Data will be made available by PDF files or other non-editable formats.

REFERENCES:
- [Background] Oteo-Alvaro A, Marin MT, Matas JA, Vaquero J. [Spanish validation of the Boston Carpal Tunnel Questionnaire]. Med Clin (Barc). 2016 Mar 18;146(6):247-53. doi: 10.1016/j.medcli.2015.10.013. Epub 2015 Dec 10. Spanish. PMID 26683079
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Fuson RL, Sherman M, Van Vleet J, Wendt T. The conduct of orthopaedic clinical trials. J Bone Joint Surg Am. 1997 Jul;79(7):1089-98. doi: 10.2106/00004623-199707000-00019. No abstract available. PMID 9234889
- [Background] Zhang L, Yang T, Pang L, Li Y, Li T, Zhang C, Yao L, Li R, Tang X. Effects of Extracorporeal Shock Wave Therapy in Patients with Mild-to-Moderate Carpal Tunnel Syndrome: An Updated Systematic Review with Meta-Analysis. J Clin Med. 2023 Nov 28;12(23):7363. doi: 10.3390/jcm12237363. PMID 38068415
- [Background] Zhang H, Zhao W, Jiang M, Song Y. Study on the effect, safety, prognosis quality and application value of extracorporeal shock wave based neural activity in carpal tunnel syndrome patients. BMC Musculoskelet Disord. 2023 Mar 13;24(1):186. doi: 10.1186/s12891-023-06285-1. PMID 36915105
- [Background] Menekseoglu AK, Korkmaz MD, Segmen H. Clinical and electrophysiological efficacy of extracorporeal shock-wave therapy in carpal tunnel syndrome: a placebo-controlled, double-blind clinical trial. Rev Assoc Med Bras (1992). 2023 Feb 17;69(1):124-130. doi: 10.1590/1806-9282.20220943. eCollection 2023. PMID 36820719
- [Background] Habibzadeh A, Mousavi-Khatir R, Saadat P, Javadian Y. The effect of radial shockwave on the median nerve pathway in patients with mild-to-moderate carpal tunnel syndrome: a randomized clinical trial. J Orthop Surg Res. 2022 Jan 25;17(1):46. doi: 10.1186/s13018-022-02941-9. PMID 35078486
- [Background] Chen KT, Chen YP, Kuo YJ, Chiang MH. Extracorporeal Shock Wave Therapy Provides Limited Therapeutic Effects on Carpal Tunnel Syndrome: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2022 May 19;58(5):677. doi: 10.3390/medicina58050677. PMID 35630095
- [Background] Tornese D, Mattei E, Lucchesi G, Bandi M, Ricci G, Melegati G. Comparison of two extracorporeal shock wave therapy techniques for the treatment of painful subcalcaneal spur. A randomized controlled study. Clin Rehabil. 2008 Sep;22(9):780-7. doi: 10.1177/0269215508092819. PMID 18728131
- [Background] Zhang YF, Liu Y, Chou SW, Weng H. Dose-related effects of radial extracorporeal shock wave therapy for knee osteoarthritis: A randomized controlled trial. J Rehabil Med. 2021 Jan 13;53(1):jrm00144. doi: 10.2340/16501977-2782. PMID 33367924
- [Background] Simplicio CL, Purita J, Murrell W, Santos GS, Dos Santos RG, Lana JFSD. Extracorporeal shock wave therapy mechanisms in musculoskeletal regenerative medicine. J Clin Orthop Trauma. 2020 May;11(Suppl 3):S309-S318. doi: 10.1016/j.jcot.2020.02.004. Epub 2020 Feb 12. PMID 32523286
- [Background] Schuh CM, Hausner T, Redl HR. A therapeutic shock propels Schwann cells to proliferate in peripheral nerve injury. Brain Circ. 2016 Jul-Sep;2(3):138-140. doi: 10.4103/2394-8108.192520. Epub 2016 Oct 18. PMID 30276290
- [Background] Guo J, Hai H, Ma Y. Application of extracorporeal shock wave therapy in nervous system diseases: A review. Front Neurol. 2022 Aug 17;13:963849. doi: 10.3389/fneur.2022.963849. eCollection 2022. PMID 36062022
- [Background] Dymarek R, Ptaszkowski K, Ptaszkowska L, Kowal M, Sopel M, Taradaj J, Rosinczuk J. Shock Waves as a Treatment Modality for Spasticity Reduction and Recovery Improvement in Post-Stroke Adults - Current Evidence and Qualitative Systematic Review. Clin Interv Aging. 2020 Jan 6;15:9-28. doi: 10.2147/CIA.S221032. eCollection 2020. PMID 32021129
- [Background] De la Corte-Rodriguez H, Roman-Belmonte JM, Rodriguez-Damiani BA, Vazquez-Sasot A, Rodriguez-Merchan EC. Extracorporeal Shock Wave Therapy for the Treatment of Musculoskeletal Pain: A Narrative Review. Healthcare (Basel). 2023 Oct 26;11(21):2830. doi: 10.3390/healthcare11212830. PMID 37957975
- [Background] Auersperg V, Trieb K. Extracorporeal shock wave therapy: an update. EFORT Open Rev. 2020 Oct 26;5(10):584-592. doi: 10.1302/2058-5241.5.190067. eCollection 2020 Oct. PMID 33204500
- [Background] Urits I, Gress K, Charipova K, Orhurhu V, Kaye AD, Viswanath O. Recent Advances in the Understanding and Management of Carpal Tunnel Syndrome: a Comprehensive Review. Curr Pain Headache Rep. 2019 Aug 1;23(10):70. doi: 10.1007/s11916-019-0811-z. PMID 31372847
- [Background] Wipperman J, Goerl K. Carpal Tunnel Syndrome: Diagnosis and Management. Am Fam Physician. 2016 Dec 15;94(12):993-999. PMID 28075090
- [Background] Zamborsky R, Kokavec M, Simko L, Bohac M. Carpal Tunnel Syndrome: Symptoms, Causes and Treatment Options. Literature Reviev. Ortop Traumatol Rehabil. 2017 Jan 26;19(1):1-8. doi: 10.5604/15093492.1232629. PMID 28436376
- [Background] Sandberg AA. A chromosomal hypothesis of oncogenesis. Cancer Genet Cytogenet. 1983 Apr;8(4):277-85. doi: 10.1016/0165-4608(83)90070-5. PMID 6831378
- [Background] Padua L, Cuccagna C, Giovannini S, Coraci D, Pelosi L, Loreti C, Bernabei R, Hobson-Webb LD. Carpal tunnel syndrome: updated evidence and new questions. Lancet Neurol. 2023 Mar;22(3):255-267. doi: 10.1016/S1474-4422(22)00432-X. Epub 2022 Dec 13. PMID 36525982
- [Background] Joshi A, Patel K, Mohamed A, Oak S, Zhang MH, Hsiung H, Zhang A, Patel UK. Carpal Tunnel Syndrome: Pathophysiology and Comprehensive Guidelines for Clinical Evaluation and Treatment. Cureus. 2022 Jul 20;14(7):e27053. doi: 10.7759/cureus.27053. eCollection 2022 Jul. PMID 36000134
- [Background] Harinesan N, Silsby M, Simon NG. Carpal tunnel syndrome. Handb Clin Neurol. 2024;201:61-88. doi: 10.1016/B978-0-323-90108-6.00005-3. PMID 38697747
- [Background] Brankack J, Klingberg F. Visual post-stimulus excitability changes in freely moving rats indicated by amplitude and peak time of evoked potentials. Acta Biol Med Ger. 1982;41(9):801-9. PMID 7164699